CLINICAL TRIAL: NCT05695560
Title: Unmet Needs of Patients Living With Von Willebrand Disease and Their Caregivers: Qualitative Survey on Current Standard of Care in Canada
Brief Title: A Survey to Describe the Experience and Unmet Needs of Persons Living With Von Willebrand Disease (VWD) and Their Caregivers
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-577-4002
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Von Willebrand Disease (VWD)
Keywords: Drug Therapy
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase 1: Adult Participants: Adult participants with severe VWD (self-bleeding assessment tool [BAT] score ≥10) and their caregivers will be enrolled as per protocol specifications. Data will be collected from participants via questionnaire, semi-structured interviews, and focus groups using a virtual platform.
  Interventions: Other: No Intervention
- Phase 2: Pediatric Participants: Pediatric participants with severe VWD (self-pediatric bleeding questionnaire [PBQ] score of ≥3 for at least one symptom and caregivers will be enrolled as per protocol specifications. Data will be collected from participants via questionnaire, semi-structured interviews, and focus groups using a virtual platform. The decision to proceed with Phase 2 will be determined following completion of Phase 1.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — As this is an observational study, no intervention will be administered.

SUMMARY:
The main aim of this study is to describe the experience and unmet needs of persons living with VWD and their caregivers in Canada.

The survey is planned to be done in two phases: The first phase will be directed at adult participants; the second phase will focus on children and teenagers. At the end of the first phase the Sponsor will decide if the second phase will be started.

Participants and their caregivers will be asked to answer a set of questions either using an online questionnaire or through interviews. The participant/caregiver's perception, experience, satisfaction, and unmet needs, and need for new treatments or new indications will be determined based on their responses to the questions.

DETAILED DESCRIPTION:
This study is a non-interventional, prospective, qualitative survey to know the unmet needs of participants living with VWD and their caregivers.

The study will enroll approximately 49 patients, taking into scope both the participant's and caregiver's perspectives, and is planned to be conducted in two phases:

Phase 1: Adult Participants Phase 2: Pediatric Participants The decision to proceed with Phase 2 will be determined at the completion of Phase 1.

This multi-center trial will be conducted in Canada. The overall time for data collection in this study is approximately 9 months.

ELIGIBILITY:
Inclusion criteria:

* Phase 1:
* Adult participants (age ≥18 years) with severe VWD (self-BAT ≥10)
* Participants who have received von Willebrand factor (VWF) treatment, either for on-demand treatment, regular prophylaxis, or situational prophylaxis (e.g., surgery) within the last 5 years
* For caregivers: Current caregiver of participants with severe VWD
* For caregivers and participants:

  * Fluent in English or French
  * Consent to participate in an individual phone interview and to fill self-administered questionnaires
  * Additional inclusion criteria for virtual focus groups:

    * Access to technology (Internet and email)
    * Consent to participate in a virtual focus group with an audio recording of the session.
* Phase 2:

  * Same as above for participants pediatric participants (age <18 years) with severe VWD (self-PBQ score of ≥3 for at least one symptom).

Exclusion criteria:

* Phase 1:
* Participants or caregivers of participants who do not have severe symptoms of VWD
* Pediatric participants (age <18 years)
* Participants who have not received any treatment (on-demand, regular or situational prophylaxis) within the last five years
* Participants who are successfully treated with desmopressin or anti-fibrinolytic medications
* Participants with inherited or acquired hemostatic or bleeding disorders other than congenital VWD (self-reported)
* Participants and caregivers of participants who show cognitive impairment (as assessed by the research nurse at the time of screening)
* Participants and caregivers who are qualified as health care practitioners currently working in a health-care capacity (e.g., physician, nurse, or healthcare aid)
* Participants or caregivers who do not reside in Canada
* Current or past participation within the last 12 months in a clinical trial
* Phase 2: Same as above excluding participants of ≥18 years of age

Ages: 0 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants and caregivers of participants diagnosed with VWD in Canada.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants Categorized Based on Bleeding Characteristics | Up to approximately 9 months
  Bleeding characteristics will include categories of bleed frequency, bleed type/location and bleed severity.
Number of Participants Categorized by Impact on Daily Life | Up to approximately 9 months
  The age-adapted impact on daily life will be categorized by questions related to quality of life, physical activity, professional life, school, financial impact, mental health, relationships, avoidance of social and physical activities, and impact on daily activities.
Number of Participants Categorized Based on Disease Management | Up to approximately 9 months
  Disease management will be categorized by need for subsequent therapies, need for additional investigations, time needed for disease management, impact on future planning and treatment access for aging participants.

SECONDARY OUTCOMES:
Time (Delay) to Treatment Initiation | Up to approximately 9 months
Duration of Therapy Schedule | Up to approximately 9 months
Number of Participants With Change in Treatment Frequency | Up to approximately 9 months
Number of Participants With Bleed Control | Up to approximately 9 months
Time to Bleed Control | Up to approximately 9 months
Number of Participants Who Missed Days at Work/School | Up to approximately 9 months
  The number of participants who missed days at work/school will include categories for patient and caregiver.
Duration of Inpatient and Outpatient Hospital Visits | Up to approximately 9 months
Participant's Experience Assessed as Number of Participants Categorized Based on Symptom Severity and Comorbidities Over Time | Up to approximately 9 months
Treatment Experience Based on Number of Participants Satisfied With the Treatment | Up to approximately 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- YolaRx Consultants, Montreal, Canada

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: NOTE: IPD Sharing Time Frame has not been entered.
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/cb2df18a41df432b?idFilter=%5B%22TAK-577-4002%22%5D